CLINICAL TRIAL: NCT03686462
Title: Virtual Reality-based Interactive Treadmill Gait Training System for Parkinson's Disease: A Randomized, Double-blind, Sham-controlled Pilot Study
Brief Title: Virtual Reality-based Interactive Treadmill Gait Training System for Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Trade, Industry & Energy(MOTIE, Korea) (Unknown)
Responsible Party: Principal Investigator, Won-Seok Kim, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1806/474-002
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Virtual Reality; Rehabilitation; Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality-based interactive treadmill training (Experimental): In this group, the subjects will receive virtual reality (VR)-based interactive treadmill training. During the 30-min training session, VR based interaction and feedback will be provided; the foot location will be visualized in the VR screen (semi-immersive condition), the obstacles will be seen in the screen from which subjects has to avoid, gait speed will be visualized, slopes of the treadmill will be changed according to the slope changes in VR and distractors will be added. Dual tasks will also be provided. Subjects in this group will receive a 30min/session, 3 sessions/week for 4 weeks, the total of 12 sessions of VR-based training.
  Interventions: Device: Virtual reality-based interactive treadmill training
- Treadmill training without VR-based interaction (Sham Comparator): The subjects in this group will receive the treadmill gait training. Virtual reality environment will be provided during the gait training but no feedback and interaction will be provided. Subjects in this group will receive a 30min/session, 3 sessions/week for 4 weeks, the total of 12 sessions of treadmill-based training.
  Interventions: Device: Treadmill training without VR-based interaction

INTERVENTIONS:
Device: Virtual reality-based interactive treadmill training — During the 30-min training session, VR based interaction and feedback will be provided; the foot location will be visualized in the VR screen (semi-immersive condition), the obstacles will be seen in the screen from which subjects has to avoid, gait speed will be visualized, slopes of the treadmill will be changed according to the slope changes in VR and distractors will be added. Dual tasks will also be provided. Subjects in this group will receive a 30min/session, 3 sessions/week for 4 weeks, the total of 12 sessions of VR-based training.
  Arms: Virtual reality-based interactive treadmill training
Device: Treadmill training without VR-based interaction — Treadmill training without VR-based interaction
  Arms: Treadmill training without VR-based interaction

SUMMARY:
Virtual-reality-based interactive treadmill system will be applied to the Parkinsons' disease patients who can walk (Hoehn and Yahr stage 2 to 4). Subjects will be randomly allocated to either VR-based treadmill training group or treadmill training without VR-based interaction. The training will be provided for 3 sessions (30min/session)/week for 4weeks, the total of 12 sessions. The outcomes will be measured at baseline, immediately after the completion of the intervention and 1 month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* definite or probable idiopathic Parkinson disease patient
* age from 18 to 80 years old
* H&Y stage 2 to 4 and who can walk 10 meter independently regardless of the use of gait aids

Exclusion Criteria:

* unstable medical conditions
* cognitive impairments which interfere with participation in virtual-reality based training
* hemispatial neglect, visual disturbance, apraxia
* other pre-existing disease involving the central nervous system (e.g. stroke, brain tumor)
* requiring the continuous manual assist with touch during the treadmill training
* can not give a consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson's disease rating scale (UPDRS) part III | Change from Baseline UPDRS III at 4 weeks
  motor domain of UPDRS, range: 0 (best) -52 (worst)

SECONDARY OUTCOMES:
10 meter walk test (10MWT) | Change from Baseline 10MWT at 4 weeks
  gait speed (m/s)
10 meter walk test (10MWT) | Change from Baseline 10MWT at 8 weeks
  gait speed (m/s)
Berg balance scale (BBS) | Change from Baseline BBS at 4 weeks
  range: 0 (worst) -52 (best)
Berg balance scale (BBS) | Change from Baseline BBS at 8 weeks
  range: 0 (worst) -52 (best)
Freezing of gait questionnaire | Change from Baseline Freezing of gait questionnaire at 4 weeks
  range: 0 (best) -24 (worst)
Freezing of gait questionnaire | Change from Baseline Freezing of gait questionnaire at 8 weeks
  range: 0 (best) -24 (worst)
Fear of falling | Change from Baseline fear of falling at 4 weeks
  Numeric rating scale ranging from 0 (no fear) to 10 (most severe fear of falling).
Fear of falling | Change from Baseline fear of falling at 8 weeks
  Numeric rating scale ranging from 0 (no fear) to 10 (most severe fear of falling).
Total number of falls during the recent 1 month | Change from Baseline total number of falls at 4 weeks
Total number of falls during the recent 1 month | Change from Baseline total number of falls at 8 weeks
User satisfaction evaluation questionnaire | At 4weeks (after the completion of whole interventions)
Gait parameters from gait analysis | Change from Baseline gait parameters at 4 weeks
  gait speed, step length, cadence
Gait parameters from gait analysis | Change from Baseline gait parameters at 8 weeks
  gait speed, step length, cadence
Unified Parkinson's disease rating scale (UPDRS) part III | Change from Baseline UPDRS III at 8 weeks
  motor domain of UPDRS, range: 0 (best) -52 (worst)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided